CLINICAL TRIAL: NCT02083081
Title: Community Intervention to Reduce Tobacco Use Among Alaska Native Pregnant Women
Brief Title: Community Intervention to Reduce Tobacco Use in Pregnant Women
Acronym: Sisters
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: Yukon Kuskokwim Health Corporation (Other); University of Minnesota (Other); National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Christi Patten, PI, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 13-008824; 1R01CA164533 (NIH)
Record Dates: First submitted 2014-03-05; First posted 2014-03-11 (Estimated); Results first posted 2022-06-28 (Actual); Last update posted 2022-06-28 (Actual); Status verified 2022-06

CONDITIONS: Nicotine Dependence
Keywords: tobacco; smoking
MeSH Terms: conditions — Tobacco Use Disorder; Smoking

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- community intervention (Experimental): Community level intervention (Social marketing campaign delivered to entire village) plus individual peer counseling sessions for enrolled pregnant women
  Interventions: Behavioral: Community level intervention
- usual care (No Intervention): Usual care provided by health aides to pregnant women

INTERVENTIONS:
Behavioral: Community level intervention — Community intervention plus individual counseling
  Arms: community intervention

SUMMARY:
In the southwest region of Alaska where the project takes place, 79% of Alaska Native women smoke cigarettes or use smokeless tobacco (ST) during pregnancy. In addition, pregnancy appears to be a high risk period for initiation of tobacco use, primarily ST, among women reporting no use of tobacco 3 months before pregnancy. Intervention efforts targeting the entire community, not only pregnant women, to address social norms about tobacco use may be effective. Thus, the investigators will evaluate the efficacy of a novel, multi-component, theory-based intervention for reducing tobacco use during pregnancy, incorporating both individually targeted and community level components delivered by female elders "Native Sisters." The intervention builds on effective community and individual-based approaches for tobacco cessation and lay health advisor approaches for cancer prevention among Native American women. As part of the intervention, a social marketing campaign including digital stories and other small media will be developed with community feedback. Individually targeted components will be six 30-40 minute telephone or home-based peer counseling sessions with pregnant women.

DETAILED DESCRIPTION:
The project will be conducted in two phases. In Phase I, the investigators will develop the social marketing components by obtaining qualitative feedback from pregnant women, family members and elders on message content and delivery channels. In Phase II, the investigators will evaluate the intervention using a group-randomized design with village as the unit of assignment. Sixteen villages will be randomly assigned to receive the intervention or control condition (usual care), with > 20 pregnant women enrolled from each village. Assessments will be completed by enrolled women through 6 months postpartum. All aspects of the project will be guided by a Community Advisory Committee.

The Specific Aims are:

Aim 1. To develop and pre-test the social marketing campaign messages and delivery channels through focus groups and individual interviews of pregnant women, family members, and elders. The focus group work will assess reasons for initiating or continuing tobacco use during pregnancy and the potential role of other community members in addressing tobacco use in pregnancy. Findings will be used to develop campaign messages and media that will be pre-tested through individual interviews and refined. Session content for the individually targeted intervention components will also be developed to align with the campaign messages.

Aim 2. To evaluate the efficacy of the intervention compared with the control condition on the biochemically confirmed 7-day point prevalence tobacco use rate at week 36 gestation and at 6 months postpartum.

Hypothesis: Compared with the control condition, the intervention will be associated with significantly lower rates of tobacco use in late pregnancy (80% vs. 65%) and at 6 months postpartum (70% vs. 55%).

Aim 3. To examine the effect of the intervention on proposed social cognitive-theory based mediators of change including perceived social norms about tobacco use and self-efficacy for non-tobacco use.

Hypothesis: Intervention effects on tobacco use at week 36 gestation and at 6 months postpartum will be mediated by perceived self-efficacy and anti-tobacco norms.

ELIGIBILITY:
Inclusion Criteria:

* Alaska Native
* >18 years of age
* able to provide written informed consent
* currently pregnant and at < 26 weeks gestation
* has access to a working telephone.

Exclusion Criteria:

* plans to have an abortion

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 352 (Actual)
Dates: Start 2014-05 (Actual); Primary Completion 2020-12 (Actual); Study Completion 2020-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christi A Patten, PhD, Principal Investigator — Mayo Clinic
Locations (1):
- Yukon Kuskokwim Health Corporation, Bethel, Alaska, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Community Intervention | Usual Care
Started | 188 | 164
Completed | 157 | 155
Not Completed | 31 | 9
Not completed — Lost to Follow-up | 31 | 9

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Community Intervention | Usual Care | Total
Number analyzed (Participants) | 188 | 164 | 352
Age, Continuous [Mean (Standard Deviation); unit: years] | 25.9 (5.0) | 25.8 (5.0) | 25.8 (5.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 188 | 164 | 352
  Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 188 | 164 | 352
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
gestational age, weeks [Mean (Standard Deviation); unit: weeks] | 27.3 (9.5) | 26.2 (10.1) | 26.8 (9.8)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Tobacco Abstinence at 6-months Post-partum
Description: Total number of participants to have biochemically confirmed tobacco abstinence at 6-months post-partum
Time Frame: 6 months postpartum
Measure: Count of Participants; unit: Participants
Arm/Group | Community Intervention | Usual Care
Number analyzed (Participants) | 188 | 164
Participants | 161 | 135
Statistical Analysis 1: Comparison: Community Intervention vs Usual Care; Test type: Superiority; p = 0.38, generalized estimating equations (GEE)

2. Primary Outcome: Number of Participants With Tobacco Abstinence at End of Pregnancy
Description: Total number of participants to have biochemically confirmed tobacco abstinence at end of pregnancy (delivery).
Time Frame: Approximately 9 months
Measure: Count of Participants; unit: Participants
Arm/Group | Community Intervention | Usual Care
Number analyzed (Participants) | 188 | 164
Participants | 122 | 111
Statistical Analysis 1: Comparison: Community Intervention vs Usual Care; Test type: Superiority; p = 0.45, generalized estimating equations (GEE)

3. Secondary Outcome: Change in Self-efficacy for Non-tobacco Use Scores
Description: Change from baseline in self-efficacy for non-tobacco use scores measured by the self-reported Smoking Confidence Questionnaire. Total scores range from 0-30, higher scores indicate better outcome.
Time Frame: Baseline, 6 months postpartum
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Community Intervention | Usual Care
Number analyzed (Participants) | 156 | 153
score on a scale | 7.2 (2.7) | 7.5 (2.6)
Statistical Analysis 1: Comparison: Community Intervention vs Usual Care; Test type: Superiority; p = 0.96, generalized estimating equations (GEE)

ADVERSE EVENTS:
Time Frame: Adverse events were collected from baseline to end of study participation for a total of approximately 15 months on all participants
Arm/Group | Community Intervention | Usual Care
All-Cause Mortality (participants affected / at risk) | 0/188 | 0/164
Serious Adverse Events (participants affected / at risk) | 0/188 | 0/164
Other Adverse Events (participants affected / at risk) | 0/188 | 0/164

LIMITATIONS AND CAVEATS:
challenges obtaining biochemical verification by mail

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-04-18): https://cdn.clinicaltrials.gov/large-docs/81/NCT02083081/Prot_SAP_000.pdf
  • Informed Consent Form (2017-03-01): https://cdn.clinicaltrials.gov/large-docs/81/NCT02083081/ICF_001.pdf